CLINICAL TRIAL: NCT02772198
Title: A Phase 1 / 2 Single Arm Study of T-cells Expressing Anti-CD19 Chimeric Antigen Receptor in Pediatric and Young Adult Patients With B-cell Malignancies
Brief Title: T-cells Expressing Anti-CD19 CAR in Pediatric and Young Adults With B-cell Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-15-2076-AT-CTIL
Record Dates: First submitted 2016-05-09; First posted 2016-05-13 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Acute Lymphoblastic Leukemia, B-precursor; Non-Hodgkin Lymphoma, B-cell
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): All patients will be treated on this single arm
  Interventions: Biological: CD19 CAR T cells

INTERVENTIONS:
Biological: CD19 CAR T cells — Autologous T cells activated and transduced with a chimeric antigen receptor targeting CD19

SUMMARY:
This phase 1 / 2 study will evaluate the response of B-cell malignancies expressing CD19 to autologous T cells transduced with a second generation anti-CD19 chimeric antigen receptor in children and young adults.

DETAILED DESCRIPTION:
Autologous T cells transduced with chimeric antigen receptors (CAR) that recognize the CD19 antigen (CD19-CAR T cells) have been used in multiple clinical trials at several institutions worldwide. We established an in-house manufacturing process for CD19-CAR T cells with a CD28 (cluster of differentiation 28) costimulatory domain.

Primary Objectives:

1. To study the safety of administration of CAR T cell at the Sheba Medical Center
2. To determine the feasibility and efficacy of administering anti-CD19-CAR T cells in children and young adults with B cell malignancies.

Secondary Objectives

1. To study in vivo and in vitro behavior of CAR T cell in patients, including persistence, expansion, cytotoxic potential and exhaustion.
2. To study the cytokine milieu in CAR treated patients.

Eligibility Patients 1-50 years of age, with a CD19-expressing B-cell malignancy that has recurred after, or not responded to, one or more standard chemotherapy-containing regimens.

Design Peripheral blood mononuclear cells (PBMCs)will be obtained by leukapheresis. Anti-CD19 CAR T cells will be manufactured from fresh autologous PBMCs. PBMC will be cultured in the presence of anti-CD3 (cluster of differentiation 3) antibody and interleukin-2 followed by retroviral vector supernatant containing the anti-CD19 CAR. Total culture time is between 7-10 days. Patients will receive lymphodepleting chemotherapy composed of cyclophosphamide and fludarabine prior to cell infusion, and on day 0 will receive one million CAR T cells per kilogram. Patients will be monitored for toxicity including cytokine release syndrome, hematologic toxicities and B-cell aplasia; for response of their underlying malignancy; and for CAR-T cell persistence in the blood, marrow and cerebral spinal fluid (CSF).

ELIGIBILITY:
Inclusion Criteria:

* Patient with relapsed or refractory B-cell malignancy
* Age 1-50 years
* CD19 expression shown by flow cytometry or immunohistochemistry on at least 70% of leukemic blasts / lymphoma cells
* Adequate CD3 count (above 250 CD3+ cells per microliter blood)
* Clinical performance status: Patients > 10 years of age: Karnofsky ≥ 50%; Patients ≤ 10 years of age: Lansky scale ≥ 50%. Exception for neurologic symptoms (e.g. paralysis) that are explained by the malignancy.
* Females of child-bearing potential must have a negative pregnancy test
* Cardiac function: Left ventricular ejection fraction >45% or shortening fraction >28%
* For patients following allogeneic bone marrow transplantation - at least 100 days post BMT with no signs or symptoms of active graft-versus-host disease.

Key Exclusion Criteria:

* Hyperleukocytosis (WBC>50,000) or rapidly progressive disease
* Pregnant or breast-feeding females
* Hepatic dysfunction, defined as bilirubin > x2 upper normal limit (except when explained by hemolysis or Gilbert) or serum glutamate oxaloacetate transaminase > x25 upper normal limit.
* Hepatitis B, Hepatitis C or HIV infection.
* Anti-neoplastic treatment given in the 2 weeks prior to apheresis, with the exception of intrathecal chemotherapy.
* Active immunosuppressive therapy

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment related adverse events as assessed by CTCAE v4. | 2 years
Overall Response Rate | 28 days
  Overall response rate = complete response (CR) + partial response (PR) + complete response with incomplete count recovery (CRi) in leukemia patients; Assessment using bone marrow evaluation for patients with leukemia, and imaging (CT / PET CT) for patients with lymphoma
Feasibility of CD19 CAR T cell production as defined by number of products successfully meeting release criteria | 12 days
  For each participant, the feasibility of generating sufficient autologous CAR T cells within 12 days will be evaluated.

SECONDARY OUTCOMES:
CAR T cell persistence as measured by enumeration of CAR T cells in the blood and bone marrow of participants | 1 year
  Enumeration of CAR T cells in the blood and bone marrow of participants
T cell activity and exhaustion profile as measured by flow cytometry | 3 months
  Assessment of T cells from peripheral blood by flow cytometry for expression of activation and exhaustion markers.
Cytokine levels in the peripheral blood of the patients | 30 days
  Measurement of cytokines in the blood of participants following CAR T cell administration

CONTACTS AND LOCATIONS:
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Itzhaki O, Jacoby E, Nissani A, Levi M, Nagler A, Kubi A, Brezinger K, Brayer H, Zeltzer LA, Rozenbaum M, Vernitsky H, Markel G, Toren A, Avigdor A, Schachter J, Besser MJ. Head-to-head comparison of in-house produced CD19 CAR-T cell in ALL and NHL patients. J Immunother Cancer. 2020 Mar;8(1):e000148. doi: 10.1136/jitc-2019-000148. PMID 32152221
- [Background] Fried S, Avigdor A, Bielorai B, Meir A, Besser MJ, Schachter J, Shimoni A, Nagler A, Toren A, Jacoby E. Early and late hematologic toxicity following CD19 CAR-T cells. Bone Marrow Transplant. 2019 Oct;54(10):1643-1650. doi: 10.1038/s41409-019-0487-3. Epub 2019 Feb 26. PMID 30809033
- [Result] Jacoby E, Bielorai B, Avigdor A, Itzhaki O, Hutt D, Nussboim V, Meir A, Kubi A, Levy M, Zikich D, Zeltzer LA, Brezinger K, Schachter J, Nagler A, Besser MJ, Toren A. Locally produced CD19 CAR T cells leading to clinical remissions in medullary and extramedullary relapsed acute lymphoblastic leukemia. Am J Hematol. 2018 Dec;93(12):1485-1492. doi: 10.1002/ajh.25274. Epub 2018 Sep 26. PMID 30187944
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Nissani A, Lev-Ari S, Meirson T, Jacoby E, Asher N, Ben-Betzalel G, Itzhaki O, Shapira-Frommer R, Schachter J, Markel G, Besser MJ. Comparison of non-myeloablative lymphodepleting preconditioning regimens in patients undergoing adoptive T cell therapy. J Immunother Cancer. 2021 May;9(5):e001743. doi: 10.1136/jitc-2020-001743. PMID 33990415